CLINICAL TRIAL: NCT02578472
Title: A Double-blind, Randomized, Controlled, 3-way Crossover, Pilot Study to Evaluate the Duration of Effects on Simulated Car Driving and Cognitive Performance After a Single Dose of JNJ-42847922, Zolpidem and Placebo in Healthy Subjects
Brief Title: Pilot Study to Evaluate the Duration of Effects on Simulated Car Driving and Cognitive Performance After a Single Dose of JNJ-42847922, Zolpidem and Placebo in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108056; 42847922EDI1011 (Other: Janssen-Cilag International NV); 2015-004203-24 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42847922; zolpidem; Placebo
MeSH Terms: interventions — seltorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Sequence ABC) (Experimental): Participants will receive Treatment A (2 capsules of 20 milligram [mg] JNJ-42847922) in Period 1, Treatment B (10 mg zolpidem and 1 placebo capsule) in Period 2 and Treatment C (2 placebo capsules) in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 2 and 6 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo
- Group 2 (Sequence BCA) (Experimental): Participants will receive Treatment B in Period 1, Treatment C in Period 2 and Treatment A in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 2 and 6 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo
- Group 3 (Sequence CAB) (Experimental): Participants will receive Treatment C in Period 1, Treatment A in Period 2 and Treatment B in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 2 and 6 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo
- Group 4 (Sequence ABC) (Experimental): Participants will receive Treatment A in Period 1, Treatment B in Period 2 and Treatment C in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 4 and 8 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo
- Group 5 (Sequence BCA) (Experimental): Participants will receive Treatment B in Period 1, Treatment C in Period 2 and Treatment A in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 4 and 8 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo
- Group 6 (Sequence CAB) (Experimental): Participants will receive Treatment C in Period 1, Treatment A in Period 2 and Treatment B in Period 3 with a washout interval of at least 3 days between treatment periods. Participants randomized to this group will be assessed for pharmacodynamic testing at 4 and 8 hours after dosing.
  Interventions: Drug: JNJ-42847922; Drug: Zolpidem; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922 — JNJ-42847922 will be administered as 40 milligram oral capsule (2 capsule*20 mg) in one of the treatment periods.
Drug: Zolpidem — Zolpidem will be administered as 1 capsule containing 10 mg in one of the treatment periods.
Drug: Placebo — Matching Placebo will be administered orally.

SUMMARY:
The purpose of the study is to evaluate the effects of JNJ-42847922, compared to zolpidem and placebo, on driving performance as assessed by the mean difference of standard deviation of lateral position (SDLP) after forced awakening using a validated driving simulator test at 2, 4, 6 and 8 hours post-evening dose.

DETAILED DESCRIPTION:
This is a single center, double-blind (neither Investigator nor participant knows which treatment the participant receives), randomized (study drug assigned by chance), 3-way cross-over (the same medications provided to all participants but in different sequence), pilot study in healthy male and female participants. Participants will be randomly assigned to 1 of 6 treatment and planning sequences. The study will consist of 3 parts: Screening Phase (between 21 days and 1 day prior to the first dose administration), a 3-way crossover double-blind, single dose treatment Phase and follow-up Phase (7 to 10 days after last dose administration). The maximum study duration for each participant will not exceed 7 weeks. The double-blind crossover treatment phase will consist of 3 treatment periods separated by a washout period of at least 3 days between dosing. Participants will receive either Treatment A (2 capsules of 20 milligram [mg] JNJ-42847922), Treatment B (10 mg zolpidem and 1 placebo capsule) or Treatment C (2 placebo capsules) in each treatment period. Driving performance will be assessed primarily by the mean difference of standard deviation of lateral position (SDLP) from an on road driving test. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) (weight [kg]/height^2[m^2]) between 18 and 30 kg/m^2 (inclusive)
* Men who are sexually active with a woman of childbearing potential must agree to use a condom, and all men must not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, for men who have not had a vasectomy, their female partners should also use an appropriate method of birth control for at least the same duration
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test pre-dose on Day 1 of each period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 3 months after receiving the last dose of study drug
* Participant has a valid driving license for more than 3 years, has driven at least 5000 kilometer (km) in the past year and is driving a car regularly
* Women of childbearing potential must practice a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies (that is, one that results in a less than 1 percent per year failure rate when used consistently and correctly)

Exclusion Criteria:

* Participant has clinically significant liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic (including cataplexy and cognitive impairment), hematologic, rheumatologic, psychiatric, or metabolic disturbances. A significant primary sleep disorder is exclusionary
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Subject has a history of substance or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 6 months before screening or positive test result(s) for alcohol and/or drugs of abuse (opiates [including methadone], cocaine, amphetamines, methamphetamines, cannabinoids, barbiturates, ecstasy and benzodiazepines) at screening or admission on Day 1 of each study period
* Current suicidal or homicidal ideation/intent/behavior
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV) or Human immunodeficiency virus (HIV) antibodies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) Assessed From an On-road Driving Test | up to 8 hours post-dose
  The SDLP will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.

SECONDARY OUTCOMES:
Mean Lateral Position (MLP) Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  The MLP will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.
Distance-keeping Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  Distance-keeping will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.
Mean Speed (MS) Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  The MS will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.
Standard Deviation of Speed (SDS) Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  The SDS will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.
Number of Head movements Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  Number of head movements will be measured from a simulated road tracking test over about 15 minutes. Instructed speed is 100 kilometer (km)/hour.
Reaction-time Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  Reaction-time will be assessed by 10 minutes of special and unexpected traffic events.
Inhibition-time Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  Inhibition-time will be assessed by 10 minutes of special and unexpected traffic events.
Alertness-time Assessed From an On-road Driving Test | 2 to 8 hours post-dose
  Alertness-time will be assessed by 10 minutes of special and unexpected traffic events.
Drive safety Score (DSS) | 2 to 8 hours post-dose
  The DSS is a composite score of driving simulator behavior ranging from 0-10, related to actual driving performance.
Subjective assessment of driving performance using visual analog scale | 2 to 8 hours post-dose
  Participants indicated the perceived quality of their driving performance on a visual analog scale, which ranged from 0 ('I drove exceptionally poorly') to 20 ('I drove exceptionally well') around a midpoint of 'I drove normally'.
Computerized Cognitive Test Battery: Detection (DET) Test | 2 to 8 hours post-dose
  Simple reaction time task measuring processing speed; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: Identification (IDN) Test | 2 to 8 hours post-dose
  Choice reaction time paradigm measuring attention; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: One Back (OBK) Test | 2 to 8 hours post-dose
  Working memory measure; mean of the log10 transformed reaction times for correct responses (lower score = better performance).
Computerized Cognitive Test Battery: One card learning | 2 to 8 hours post-dose
  A visual recall test scored using arcsine transformation of the proportion of correct responses.
Computerized Cognitive Test Battery: Trailmaking Test Form B (TMT-B) | 2 to 8 hours post-dose
  TMT-B is a paper-and-pencil measure of divided attention and executive function (tracking, sequencing). The participant is instructed do draw a line to connect a set of 25 consecutively numbered and lettered circles, alternating sequentially between numbers and letters. The participant is instructed to work as quickly as possible while still maintaining accuracy. The test requires approximately 2 minutes to complete, alternate forms are available. Scores include time to completion and errors.
Postural Stability Test | 2 to 8 hours post-dose
  Postural stability will be measured by body sway meter which allows measurement of body movements in a single plane. Body sway is measured with a pot string meter (celesco) based on the Wright ataxiameter (Wright, 1971). With a string attached to the waist, all body movements over a period of time are integrated and expressed as millimeter sway. The total period of body sway measurement will be two minutes.
Karolinska Sleepiness Scale (KSS) Score | 2 to 8 hours post-dose
  The KSS is a participant-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep).
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to Follow-up (7-10 days after last dose of study drug)
  An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Relationship between duration of changes in driving ability and plasma concentrations of JNJ-42847922 | Pre-dose and Day 1 post-dose
  Relationship between duration of changes in driving ability and plasma concentrations of JNJ-42847922 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Leiden, Netherlands